CLINICAL TRIAL: NCT05452122
Title: Decoding and Selective Modulation of Human Memory During Awake/Sleep Cycles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Iowa (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Itzhak Fried, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: U01NS123128 (NIH); 1U01NS123128-01 (NIH)
Record Dates: First submitted 2022-06-18; First posted 2022-07-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Memory, Delayed
Keywords: sleep; stimulation; memory; learning; single-unit
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Auditory and Electrical Stimulation — Electrical and auditory stimulation will be applied during sleep.

SUMMARY:
The proposed project seeks to elucidate memory processes and consolidation during sleep by leveraging the unique capability of direct recordings from the human brain at multiple levels of resolution-single neurons, localized neuronal assemblies, intracranial local field potentials-during rich behavioral tasks with real-life narratives and extracting neural features that relate to different aspects of episodic experience. The investigators will further probe causal mechanisms of consolidation by application of auditory and electrical stimulations during sleep and its effect on modulating memory processes.

ELIGIBILITY:
Inclusion Criteria:

* All epilepsy patients between the ages of 18 and 65 who undergo depth electrode placement for clinical purposes
* Eligibility is determined by the epilepsy surgery team (based on neuropsychological testing and on psychiatric evaluation)
* Willing to provide informed consent and participate the study

Exclusion Criteria:

* Neurological or psychiatric issues, other than epilepsy, that would put the patient at risk
* Patient is younger than 18 or older than 65 years of age
* Unwilling to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Recognition Accuracy | 1-2 days contained within the participants' 1-2 week hospital stay; Specifically for each experiment, the outcome measure will be computed during the pre- and post-sleep memory tasks
  Accuracy will be analyzed to evaluate performance on memory tasks before and after sleep, specifically the ability to recognize correct items compared to all items. Accuracy will be measured using the sum of true positive and true negative divided by the total number of items. A within-subjects design will be employed and accuracy for stimulated vs. non-stimulated items will be compared.
Recognition Discriminability (D-prime) | 1-2 days contained within the participants' 1-2 week hospital stay; Specifically for each experiment, the outcome measure will be computed during the pre- and post-sleep memory tasks.
  Discriminability will be analyzed to evaluate performance on memory tasks before and after sleep, specifically the ability to recognize target items from distractor items. Discriminability will be measured using a discriminability index (d-prime). In addition to d-prime being a normalized metric, it provides critical and complementary information to the accuracy metric (Outcome 1) given that it is a measure of sensitivity (and not bias) in the cases where data labels are not balanced . A within-subjects design will be employed and discriminability for stimulated vs. non-stimulated items will be compared.

SECONDARY OUTCOMES:
Power sleep oscillations | 1-2 days contained within the participants' 1-2 week hospital stay. Specifically for each experiment, the outcome measure will be computed during the sleep period between pre and post-sleep memory tasks.
  The power of slow waves, spindles, ripples (all in units of dbm) will be computed. Employing a within-subjects design, the investigators will compare the change in the power of these oscillatory features for stimulated vs. non-stimulated items.
Neuronal replay index | 1-2 days contained within the participants' 1-2 week hospital stay. Specifically for each experiment, the outcome measure will be computed during the sleep period between pre and post-sleep memory tasks.
  Neuronal replay index, defined as the percentage of time during which neurons manifest replay-like activation as compared to the duration of deep sleep will be computed. Employing a within-subjects design, the investigators will compare the replay measure for stimulated vs. non-stimulated items.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make data available in accordance with the latest BRAIN Initiative Data Sharing Plan. The data consists of intracranial recordings from human epilepsy patients while participants perform a cognitive task during awake periods and follow-up recordings during overnight sleep or nap sessions. These datasets will be shared in a HIPAA-compliant manner (anonymized and coded) and will not include any sensitive information such as Protected Health Information. The investigators plan to deposit the data using the NIH Data Archive Brain Initiative platform, specialized at storage and organization of invasive neurophysiology data.
Supporting Information: Analytic Code
Time Frame: All data will be provided by the time publication occurs or per NIH latest policies for the data to be shared periodically via specialized storage for invasive neurophysiology data.
Access Criteria: Researchers can request access to the data under collaborative and co-authorship agreements prior to the end of the funding period or before publication.
URL: https://dabi.loni.usc.edu/home